CLINICAL TRIAL: NCT04527900
Title: The "Upproach" Approach: A Phase 2 Study Of Upfront Intensity Modulated Proton Beam Therapy (Impt) And Concurrent Chemotherapy For Post-Operative Treatment In Loco-Regionally Advanced Endometrial Cancer
Brief Title: The UPPROACH (Upfront Intensity Modulated Proton Beam Therapy) Approach
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: SOC changed and low enrollment
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00092397
Record Dates: First submitted 2020-08-14; First posted 2020-08-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Gynecologic cancers; Radiotherapy; Proton Therapy; Chemotherapy; Chemoradiation
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Concurrent chemoradiation (Experimental): Concurrent carboplatin and paclitaxel and IMPT (Intensity Modulated Proton Therapy)
  Interventions: Drug: carboplatin and paclitaxel; Radiation: pelvic IMPT (Intensity Modulated Proton Therapy)

INTERVENTIONS:
Drug: carboplatin and paclitaxel — carboplatin and paclitaxel 5-6 cycles (dosage per standard of care according to treating oncologist)
Radiation: pelvic IMPT (Intensity Modulated Proton Therapy) — whole pelvis will receive a total dose of 4500 cGy in 25 fractions to 5040 cGy in 28 fractions

SUMMARY:
A phase 2 study with the primary objective of testing treatment compliance of Upfront Intensity Modulated Proton Beam Therapy (IMPT) and Concurrent Chemotherapy (UPPROACH) for Post-operative Treatment in Loco-regionally Advanced Endometrial Cancer is non-inferior to the historic compliance rate of the chemoradiation arm of GOG 258 study

DETAILED DESCRIPTION:
While there is a consensus that both adjuvant ChT and RT benefit patients with respect to locoregional and distant control, the sequencing of these therapies varies between institutions. Common approaches include sequential treatment, with 4-6 cycles of ChT followed by RT, sandwich therapy with RT sandwiched between 3 cycles of ChT, or concurrent CRT. Small retrospective studies have shown a benefit with respect to PFS and OS in the sandwich approach, however this has not been replicated in larger studies.

In more recent years, proton beam therapy (PBT) has become an increasingly common modality for the treatment of uterine malignancies and is capable of even more precise dose distributions than photon-based RT due to intrinsic properties of these much heavier particles. Dosimetric/planning studies from other institutions confirm the significant reduction of dose to critical normal tissues like bladder, bowel, rectum, and bone marrow.

Preliminary data from the University of Maryland Medical Center has suggested that IMPT using pencil beam scanning is feasible in patients with endometrial cancer, with only 10% of patients developing grade 2 GI toxicity and no patients developing ≥ grade 3 GI or GU toxicities (abstract under review).

The investigators would like to test the hypothesis that in the postoperative setting, patients with advanced endometrial cancer will be able to complete a course of full dose ChT - carboplatin and paclitaxel - concurrent with upfront pelvic IMPT.

ELIGIBILITY:
Inclusion Criteria:

1. Surgery must have included a hysterectomy. Bilateral salpingo-oophorectomy, pelvic lymph node sampling, para-aortic lymph node sampling, and omentectomy are optional
2. Patients will be staged according to FIGO 2009 staging system. Eligibility is defined based on clinical-pathologic features.
3. Patients with endometrioid endometrial cancer with the following:

   * Stage IA grade 3 with extensive LVSI
   * Stage IB grade 3
   * Stage II
   * Stage III (A, B, and C)
   * Stage IVA who are recommended adjuvant whole pelvic RT (+/- lower para-aortic up to renal hilum) and systemic chemotherapy.
4. Patients with clear cell, serous papillary carcinoma, or carcinosarcoma with stages IA-III who are recommended adjuvant whole pelvic RT (+/- lower para-aortic up to renal hilum) and systemic chemotherapy.
5. Patients with a GOG Performance Status of 0, 1, or 2
6. Patients with adequate organ function, reflected by the following parameters:

   * WBC ≥ 3000/mcl
   * Absolute neutrophil count (ANC) ≥ 1000/mcl
   * Platelet count ≥ 100,000/mcl
   * SGOT, SGPT, and alkaline phosphatase ≤ 2.5 X upper limit of normal (ULN)
   * Bilirubin ≤ 1.5 X ULN
   * Creatinine ≤ institutional ULN (if serum creatinine > ULN, estimated GFR ≥ 45 ml/min)
7. Patients who have signed an approved informed consent and authorization permitting release of personal health information
8. Patients must be 18 years of age or older

Exclusion Criteria:

1. Patients with leiomyosarcoma
2. Patients with clinically significant pelvic or para-aortic nodal disease, on post-surgery CT scan, that was not dissected and would require higher boost dose
3. Patients with recurrent endometrial cancer with gross nodal or vaginal disease requiring high dose radiotherapy, or history of prior chemotherapy
4. Patients with a history of prior pelvic/abdominal RT or with history of prior cancer treatment that contraindicates this protocol therapy including history of prior chemotherapy for any other malignancy.
5. Patients with a history of serious co-morbid illness or uncontrolled illnesses that would preclude protocol therapy
6. Patients with an estimated survival of less than three months
7. Patients with FIGO 2009 Stage IVB endometrial cancer
8. Patients with a history of myocardial infarction, unstable angina, or uncontrolled arrhythmia within 3 months from enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Compliance rates | End of study, approximately 4 years
  This will be measured as proportion of patients completing full 6 cycles of chemotherapy concurrently with IMPT

SECONDARY OUTCOMES:
Acute GI and urinary toxicity | once a week during radiation treatment (5-6 weeks)
  Measured by CTCAE (Common Terminology Criteria for Adverse Events)
Acute GI and urinary toxicity | once a week during radiation treatment (5-6 weeks)
  Measured by PRO-CTCAE (Patient reported outcomes Common Terminology Criteria for Adverse Events)
Acute GI and urinary toxicity | once a week during radiation treatment (5-6 weeks)
  Measured by EPIC (Expanded Prostate Cancer Index Composite ) bowel and urinary domain
Acute hematologic toxicity | Prior to each cycle of chemotherapy (once every 21 days for 106 days)
  Measured by CTCAE (Common Terminology Criteria for Adverse Events)
Late GI and urinary toxicity | 6-month following radiation therapy
  Measured by CTCAE (Common Terminology Criteria for Adverse Events)
Late GI and urinary toxicity | 6-month following radiation therapy
  Measured by PRO-CTCAE (Patient reported outcomes Common Terminology Criteria for Adverse Events)
Late GI and urinary toxicity | 6-month following radiation therapy
  Measured by EPIC (Expanded Prostate Cancer Index Composite ) bowel and urinary domain

CONTACTS AND LOCATIONS:
Overall Officials: Pranshu Mohindra, MD, Principal Investigator — University of Maryland/Maryland Proton Treatment Center
Locations (4):
- United States (4):
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - UMMC, Baltimore, Maryland
  - Central Maryland Radiation Oncology, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland

IPD SHARING:
Plan to Share IPD: No